CLINICAL TRIAL: NCT05741593
Title: Qualitative Analysis of Interviews Between Pharmacist and Elderly Patients Treated with Antithrombotics for an Ischemic Stroke.
Acronym: QUATRO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1074; 2023-A00181-44 (Other: ID-RCB)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Qualitative study; semi-structured interview; antithrombotic; stroke; medication adherence
MeSH Terms: conditions — Stroke; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients having had a stroke: elderly patients previously treated with an antithrombotic and admitted to hospital for an ischemic stroke
  Interventions: Other: Analysis of the verbatim from the transcription of the recorded interviews.

INTERVENTIONS:
Other: Analysis of the verbatim from the transcription of the recorded interviews. — recorded semi-structured interviews between the patients and the pharmacist

SUMMARY:
Cerebrovascular accident is the 2nd leading cause of death and the leading cause of disability in the world. There are brakes and levers of medication adherence in the context of secondary prevention treatment in stroke.

DETAILED DESCRIPTION:
Cerebrovascular accident is the 2nd leading cause of death and the leading cause of disability in the world. The probability of stroke recurrence is high: about 25% the first year , and 30 to 40% in the 5 years following the stroke. Recurrent strokes are responsible for significant disability, institutionalization, major neurocognitive disorders, and death.

In order to reduce the risk of stroke recurrence, multiple secondary prevention strategies have demonstrated their effectiveness, such as the prescription of drugs (in particular statins and antithrombotics), the establishment of a balanced diet, the practice of an activity physical, or even tobacco addiction.

However, the effectiveness of these strategies is optimal if and only if patients adhere to them.

In addition, previous studies have focused on the brakes and levers of medication adherence in the context of secondary prevention treatment in stroke.

In elderly patients, other obstacles could have been identified by specific studies, such as cognitive, sensory, functional disorders or even isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and over
* Patients hospitalized for an ischemic stroke or a recurrence of ischemic stroke, already being treated with an antithrombotic treatment (antiplatelet agent or anticoagulant ) prior to the stroke
* Patients living at home and with a plan to return home.
* Patients who did not object to the study and who gave their consent for the recording of the interview

Exclusion Criteria:

* Patients with cognitive disorders or stroke sequelae that do not allow a semi-directive interview to be carried out (at medical discretion).
* Non-French speaking patients

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 and over, hospitalized for an ischemic stroke or a recurrence of ischemic stroke, being already treated with an antithrombotic treatment hospitalized at the Charpennes hospital with a plan to return home
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of the verbatim from the transcription of the recorded interviews. | one year
  Describing the content of discussions, relating to antithrombotic treatment for secondary prevention, between elderly patients previously treated with antithrombotics and admitted to hospital for an ischemic stroke and a pharmacist

SECONDARY OUTCOMES:
Analysis of verbatim statements from the transcription of recorded interviews on patients' representations and beliefs regarding antithrombotics | 15 to 60 minutes per patient
  Exploring patients' representations and beliefs regarding antithrombotics before and after the onset of stroke or recurrence of stroke
Analysis of verbatim statements from the transcription of recorded interviews on patients' medication adherence to antithrombotics | 15 to 60 minutes per patient
  Explore patients' medication adherence to antithrombotics before the onset of stroke or recurrence of stroke
Analysis of verbatim statements from the transcription of recorded interviews on the impact of the occurrence of stroke or recurrence of stroke on medication adherence | 15 to 60 minutes per patient
  Explore the impact of stroke occurrence or stroke recurrence on patient medication adherence (including motivation, ambivalence, confidence in medication benefits)
Analysis of verbatim statements from the transcription of recorded interviews on the obstacles and levers to medication adherence | 15 to 60 minutes per patient
  Identify the barriers and levers to drug adherence with antithrombotics

CONTACTS AND LOCATIONS:
Locations (1):
- institute of aging - Hôpital des Charpennes, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No